CLINICAL TRIAL: NCT05140603
Title: Ambispective Cohort Study to Evaluate the Effectiveness, Safety and Tolerance of a Doravirine-based Antirretroviral Regimen as a Switching Strategy in Virologically Supressed HIV Infected Patients: Real-world Data
Brief Title: Ambispective Cohort Study to Evaluate the Efficacy, Safety, and Tolerance of an Antiretroviral Regimen With Doravirine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-DOR-2021-01
Record Dates: First submitted 2021-11-16; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients who received a doravirine-based regimen.

SUMMARY:
Observational, ambispective single-center cohort study, including 150 patients who received or are receiving a doravirine-based regimen plus two NRTI or a dual therapy of doravirine plus dolutegravir (DTG) or bDRV in routinely clinical practice.

DETAILED DESCRIPTION:
Observational, ambispective single-center cohort study, including 150 patients who received or are receiving a doravirine-based regimen plus two NRTI or a dual therapy of doravirine plus dolutegravir (DTG) or bDRV in routinely clinical practice.

All patients who were switched to a doravirine-based regimen from date of its availability in the center (September 2020) due to clinical considerations and have available records will be retrospectively included until date of study approval (expected on July 2021).

Minor resistances in a basal genotype to NNRTI or previous failure to NNRTI as nevirapine or efavirenz will be accepted if doravirine it is combined with a high genetic barrier drug with complete activity.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years HIV-1 infected subjects.
* Switched to a doravirine-based ART regimen under clinician criteria.

Exclusion Criteria:

* Doravirine major resistance mutations (accessory mutations are allowed).
* Major mutations to any of the other drugs combined with doravirine.
* Pregnancy, active tuberculosis or any condition that contraindicate the use of doravirine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were switched to a doravirine-based regimen from the date of its availability in our center (September 2020) due to clinical considerations and have records available will be retrospectively included until the study approval date (expected July 2021).
  Minor resistances in a baseline genotype to NNRTI or prior failure to NNRTI such as nevirapine or efavirenz will be accepted if doravirine is combined with a fully active high genetic barrier drug.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with an HIV-1 viral load ≤ 50 and ≤ 200* copies/ml using snapshot algorithm. | Up to 96 weeks.
  FDA snapshot algorithm (ITT-exposed).

SECONDARY OUTCOMES:
Rate of changes in renal biomarkers. | Up to 48 weeks.
  Changes in renal biomarkers from baseline (mean absolute changes in glomerular filtrate estimation (eGFR and CKD-epi equation)/24 (interim analysis) and 48 weeks.
Rate of changes in hepatic parameters. | Up to 48 weeks.
  Changes in hepatic parameters from baseline (median percentage of change in ASL, AST, GGT, AF and bilirubin).
Rate of changes in lipid parameters. | Up to 48 weeks
  Changes in lipid parameters from baseline (median percentage of change in total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, CT-HDL ratio.
Tolerability rate of study patients. | Up to 48 weeks.
  Number of interactions, adverse events and toxicities.
Death rates among trial patients. | Up to 48 weeks.
  Number of patients who died during or after the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Espinosa Aguilera, Principal Investigator — Virgen del Rocío University Hospital
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain